CLINICAL TRIAL: NCT05818995
Title: Therapeutic Drug Use in Patients With Chronic Kidney Disease (CKD): a Multicenter Retrospective Real-world Study
Brief Title: Therapeutic Drug Use for CKD Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li，MD, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYX-LX-20230101
Record Dates: First submitted 2023-03-23; First posted 2023-04-19 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Diabetes nephropathy; Drug effectiveness; Drug safety; Drug economics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Dipeptidyl-Peptidase IV Inhibitors; Glucagon-Like Peptide-1 Receptor Agonists; Sodium-Glucose Transporter 2 Inhibitors; Calcium Channel Blockers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- CKD G1: GFR ≥90 mL/(min·1.73m2)
  Interventions: Drug: angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, calcium channel blockers, β Receptor blocker
- CKD G2: GFR 60~89 mL/(min·1.73m2)
  Interventions: Drug: angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, calcium channel blockers, β Receptor blocker
- CKD G3: GFR 30~59 mL/(min·1.73m2)
  Interventions: Drug: angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, calcium channel blockers, β Receptor blocker
- CKD G4: GFR 15~29 mL/(min·1.73m2)
  Interventions: Drug: angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, calcium channel blockers, β Receptor blocker
- CKD G5: GFR <15 mL/(min·1.73m2)
  Interventions: Drug: angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, calcium channel blockers, β Receptor blocker

INTERVENTIONS:
Drug: angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, calcium channel blockers, β Receptor blocker — Drug types: angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, calcium channel blockers, β Receptor blockers Treatment prescription: medication alone or in combination Dose used: <standard dose, standard dose, >standard dose Frequency of administration: once a day, twice a day, three times a day.

SUMMARY:
Chronic kidney disease (CKD), characterized as renal dysfunction, is recognized as a major public health problem with high morbidity and mortality worldwide. This study aimed to analyze the common drug use and combinations of different stages and types of CKD patients. The study is a multicenter retrospective study involving three hospitals. Investigators reviewed and analyzed all patients diagnosed with chronic kidney disease from July 1, 2020 to June 30, 2022. Chronic kidney disease was defined as eGFR less than 60 mL/min per 1·73 m(2) or the presence of albuminuria. The study selected seven types of drugs based on hospital electronic medical record data, including β Receptor blockers, angiotensin converting enzyme inhibitor blockers, angiotensin II receptors, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, and calcium channel blockers. Chi-square test, Mann-Whitney Wilcoxon test, and Kruskal Wallis test will be used for statistical analysis. The main purpose of this study is to provide evidence for promoting rational drug use in CKD patients by describing the drug use. The secondary purpose of the study is to explore the efficacy, safety and economy of SGLT-2 inhibitors in diabetes nephropathy (DN).

ELIGIBILITY:
Inclusion Criteria:

1. Visit time (based on admission time for inpatients) is from July 1, 2020 to June 30, 2022
2. Any diagnostic type of the patient's visit includes CKD related diagnostics
3. Age ≥ 18 years old

Exclusion Criteria:

1. Diagnosis includes malignant tumors
2. Diagnosis includes uremia, hemodialysis, or peritoneal dialysis
3. Diagnosis includes jaundice
4. Incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with chronic kidney disease from July 1, 2020 to June 30, 2022
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
eGFR | October , 2023
  The current treatment status and medication regimen of CKD patients with different risk stratification were analyzed by GFR staging.
albuminuria | October , 2023
  The current treatment status and medication regimen of CKD patients with different risk stratification were analyzed by albuminuria grading.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Li，MD, Jinan, Shandong, China